CLINICAL TRIAL: NCT05404009
Title: Prospective, Digitized Dietary Intake Monitoring in Individuals Undergoing Cancer Therapy
Brief Title: Collecting Dietary Information From People Undergoing Cancer Treatment
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 22-149
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Receiving Allogeneic Hematopoietic Cell Transplants
Keywords: Dietary Intake Monitoring; 22-149

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to develop a secure method of collecting dietary and nutritional intake information from people with cancer. The researchers will use this information to learn more about how dietary information may relate to cancer diagnosis and response to treatment, and to identify factors that may lead to higher or lower risk of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient is receiving or planning to receive therapy for cancer.
* Patient (or caregiver) has sufficient English proficiency.

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Several prospective subcohorts of patients will be recruited in a rolling fashion. The first 3 subcohorts will comprise allo-HCT, auto-HCT, and CAR-T recipients.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
establish a prospective database | 2 years
  of nutritional intake data from immunotherapy patients that can be paired with the fecal and blood biospecimens already being collected under other protocols (06-107, 16-834) for the purpose of conducting studying correlations between nutrition, gut microbiome, and clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Peled, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm